CLINICAL TRIAL: NCT02173925
Title: Ghrelin, Leptin, Serotonin, TRPV1, NGF and GDNF Expression in the Patients With Functional Dyspepsia
Brief Title: Gut Hormone, Nociceptors, Neurotrophic Factors Expression in Functional Dyspepsia
Acronym: FD
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Nayoung Kim, M.D, Ph.D., Seoul National University Bundang Hospital
Other Study IDs: B-1101/119-010
Record Dates: First submitted 2014-06-13; First posted 2014-06-25 (Estimated); Last update posted 2015-01-07 (Estimated); Status verified 2015-01

CONDITIONS: Functional Dyspepsia; H. Pylori Infection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample (plasma and serum), samples with DNA and paraffin-embedded tissue. During the endoscopic examination, one pair of biopsies was obtained from the greater curvature of high body. Biopsies are taken using standard biopsy forceps.

GROUPS / COHORTS (2):
- Functional dyspepsia group: Patients who had epigastric pain or discomfort with normal upper endoscopy and no organic evidence for explaining these symptoms
- Control group: Subjects with normal endoscopic finding who do not have any gastrointestinal symptoms

SUMMARY:
The pathophysiology of functional dyspepsia is still unclear but several peptides have been indicated in the etiological factors in FD. Ghrelin and leptin are involved in regulation of appetite and gut motility and serotonin is a typical neurotransmitter related with sensory and motor functions of gut. On the other hand, transient receptor potential vanilloid receptor 1 (TRPV1) has been proposed to be involved with functional gastrointestinal disorder, and expression of this receptor could be regulated by nerve growth factor (NGF) or glial cell-line derived neurotrophic factor (GDNF). The investigators aimed to determine whether expressions of ghrelin,leptin, serotonin,TRPV1,GDNF and NGF in blood or gastric mucosa of FD patients are different from those in healthy controls, and whether some changes of their expression correlate with certain dyspeptic symptoms. The investigators also investigated the effect of H. pylori infection by comparing their expressions before and one year after H. pylori eradication.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who completed upper GI endoscopy and questionnaire about gastrointestinal symptoms

Exclusion Criteria:

* Daily user of NSAID or anticoagulants
* with concomitant systemic diseases such as diabetes mellitus or any malignancy
* Participants with major depression, psychosis, eating disorder
* Participants with typical reflux symptom
* Patients with Benign gastric ulcer or duodenal ulcer
* Patients with past gastrointestinal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had epigastric pain or discomfort with normal upper endoscopy and no evidence for explaining these symptoms were prospectively enrolled in Seoul National University Bundang Hospital. All participants underwent esophagogastroduodenoscopy. During endoscopy, biopsies were taken from both antrum and body for histological evaluation, determining H. pylori infection status.
  Participants were divided into control and patients according to the Rome III criteria. Patients group were subclassified into 3 categories; PDS (postprandial distress syndrome), EPS(epigastric pain syndrome) or mixed (PDS+EPS)
Sampling Method: Non-Probability Sample
Enrollment: 314 (Actual)
Dates: Start 2011-02; Primary Completion 2014-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Level of fasting plasma acyl ghrelin | Baseline

SECONDARY OUTCOMES:
Change of gastric mRNA ghrelin, leptin, TRPV1, NGF and GDNF expression and blood level of acyl ghrelin, leptin and serotonin | Baseline/ 1year
Expression of gastric ghrelin, leptin, TRPV1, NGF and GDNF mRNA and blood level of des-acyl ghrelin and serotonin | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Nayoung Kim, M.D, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea